CLINICAL TRIAL: NCT07335211
Title: A Multicenter, Randomized, Single-blind, Active Controlled, Phase III Clinical Trial to Evaluate the Efficacy and Safety of HUC3-637 in Patients With Primary Open Angle Glaucoma or Ocular Hypertension
Brief Title: Efficacy and Safety of HUC3-637 in Patients With Primary Open Angle Glaucoma or Ocular Hypertension
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Huons Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUC3-637
Record Dates: First submitted 2026-01-05; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Primary Open Angle Glaucoma (POAG); Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HUC3-637 (Experimental): Dorzolamide, Timolol
  Interventions: Drug: HUC3-637
- HUC3-637-R (Active Comparator): Dorzolamide, Timolol
  Interventions: Drug: HUC3-637-R

INTERVENTIONS:
Drug: HUC3-637 — Ophthalmic solution instilled directly into the eye (topical ocular administration)
  Arms: HUC3-637
Drug: HUC3-637-R — Ophthalmic solution instilled directly into the eye (topical ocular administration)
  Arms: HUC3-637-R

SUMMARY:
A multicenter, randomized, single-blind, active controlled, phase III clinical trial to evaluate the efficacy and safety of HUC3-637 in patients with primary open angle glaucoma or ocular hypertension

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 19 years and older
* Participants diagnosed with POAG or OH
* Have fully explained and understood the study and have voluntarily given written informed consent.

Exclusion Criteria:

* Acute or chronic angle-closure glaucoma
* Congenital glaucoma, secondary glaucoma (open-angle glaucoma)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Mean change in diurnal IOP | 12 week

CONTACTS AND LOCATIONS:
Locations (1):
- Kangbuk Samsung Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No